CLINICAL TRIAL: NCT00468949
Title: Health-Related Quality of Life in Patients With Dupuytren's Disease: A Prospective Cohort Study.
Brief Title: Health-Related Quality of Life in Patients With Dupuytren's Disease
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Dr. Achilleas Thoma, McMaster University
Organization: McMaster University (Other)
Other Study IDs: 06-2713
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Dupuytren's Contracture
Keywords: Health-Related Quality of Life; Dupuytren's Disease; Health Utilities Index; Short Form-36;; Michigan Hand Outcomes Questionnaire
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients undergoing excision surgery for their dupuytren's contracture
- 2: Patients not undergoing surgery for their excision surgery

SUMMARY:
Main Research Questions:

We want to measure the change in quality of life in Dupuytren's disease patients who do and do not undergo surgery. Also, we want to test the validity of health related quality of life measurements in patients with Dupuytren's disease.

Why is this research important? Some patients with Dupuytren's contracture require excision surgery or palmar fasciectomy. Other patient's with Dupuytren's contracture do not require surgery; however, these patients may need surgery in the future. No studies have reported the health-related quality of life of patients with Dupuytren's disease whether related to surgical intervention or not.

What is being studied? We are studying the difference and change in health-related quality of life in patients suffering from Dupuytren's disease who require excision surgery and do not require surgery.

DETAILED DESCRIPTION:
Previous research on Dupuytren's disease has not reported the health-related quality of life (HRQL) of patients' whether related to surgical intervention or not. The primary objective of this study is to measure the change in HRQL in Dupuytren's contracture patients who do and do not undergo palmar fasciectomy. Health related quality of life will be measured using the 1) Health Utilities Index Mark III (HUI3); 2) Short Form-36 (SF-36); and the 3) Michigan Hand Outcomes Questionnaire (MHQ). The secondary objective is to look at the measurement properties, including the reliability and responsiveness, of each of the three HRQL instruments when they are used in patients with Dupuytren's contracture. We will also assess the concurrent validity of each of the HRQL instruments.

ELIGIBILITY:
Inclusion Criteria:

* patients who have the diagnosis of Dupuytren's disease
* able to comprehend English to complete the self-reported questionnaires
* willing to provide informed consent.

Exclusion Criteria:

* patients who have had previous Dupuytren's contracture surgery on the same hand
* patients who have carpal tunnel syndrome, rheumatoid arthritis, connective tissue disorder, tenosynovitis, or another condition that could affect quality of life
* patients who are under the age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with dupuytren's contracture
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD MSC, Principal Investigator — St. Josephs Hamilton Health Care / McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Thoma A, Kaur MN, Ignacy TA, Levis C, Martin S, Duku E, Haines T. Health-related quality of life in patients undergoing palmar fasciectomy for Dupuytren's disease. Plast Reconstr Surg. 2014 Jun;133(6):1411-1419. doi: 10.1097/PRS.0000000000000177. PMID 24569424